CLINICAL TRIAL: NCT07043868
Title: Effects and Feasibility of Photobiomodulation at 830 Nanometers in the Treatment of Diabetic Ulcers: a Randomized, Double-blind Clinical Trial
Brief Title: Effects and Feasibility of Photobiomodulation at 830nm Nanometers in the Treatment of Diabetic Ulcers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Piaui (Other)
Responsible Party: Principal Investigator, Vinicius Saura Cardoso, Principal Investigator, Federal University of Piaui
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 7.488.044
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Diabete Type 2; Diabetic Foot Ulcer; Photobiomodulation; Low Level Laser Therapy
Keywords: diabetic foot ulcer; photobiomodulation; low level laser therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Foot | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CG + conventional dressing (Active Comparator): The group will receive application of Gallium Arsenide LASER (GasAs) 904nm 10J/cm2 associated with Helianthus annuus oil dressing.
  Interventions: Device: Low Level Laser Therapy
- GL1 4J/cm2 +conventional dressing (Experimental): The group will receive application of Gallium Arsenide LASER (GasAs) 830nm 4 J/cm² associated with Helianthus annuus oil dressing.
  Interventions: Device: Low Level Laser Therapy
- GL2 8J/cm2 +conventional dressing (Experimental): The group will receive application of Gallium Arsenide LASER (GasAs) 830nm 8J/cm² associated with Helianthus annuus oil dressing.
  Interventions: Device: Low Level Laser Therapy
- GL1 12J/cm2 +conventional dressing (Experimental): The group will receive application of Gallium Arsenide LASER (GasAs) 830nm 12J/cm² associated with Helianthus annuus oil dressing.
  Interventions: Device: Low Level Laser Therapy

INTERVENTIONS:
Device: Low Level Laser Therapy — Painless, non-invasive treatment
  Other Names: Photobiomodulation

SUMMARY:
Diabetic foot ulcers (DFU) are among the late complications of DFU, defined as skin lesions that involve the dermis to deeper structures, such as muscles and bones. Although preclinical studies have demonstrated the effects of GaAs 830 nm in diabetic wounds, no clinical studies have been performed, revealing the need for more in-depth analyses to identify the effects and ideal parameterization of PBM with GaAs 830 nm wavelength in the treatment of diabetic ulcers, improving quality of life, as well as to understand the therapeutic feasibility, time required for healing and recurrence rates of these lesions. Experimental, randomized, controlled, double-blind study, with blinding applied to the evaluator and participants. A total of 136 volunteers will be recruited for the research, carried out at the Integrated Center of Medical Specialties (CIEM) - Polyclinic. LLLT GaAs 830nm will be used with three dosages of low, medium and high intensity (4 J/cm², 8 J/cm², 12 J/cm²). The study will have three intervention groups using LLLT with GaAs 830nm and a control group, in which LLLLT will be performed with a GaAs 904nm wavelength and a dose of 10 J/cm², according to Saura et al (2024). This study was approved by the local Research Ethics Committee (Opinion 7,488,044), conducted in accordance with the Declaration of Helsinki and in accordance with the CONSORT (Consolidated Standards of Reporting Trials) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of both sexes
* Age over 18 years
* Medical diagnosis of diabetes mellitus (DM)
* Presence of diabetic ulcer

Exclusion Criteria:

* Autoimmune diseases
* Infected diabetic ulcers
* Osteomyelitis
* Ischemia
* Concomitant psychiatric disorders
* Contraindications to treatment methods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-01-10 (Estimated); Study Completion 2028-01-10 (Estimated)

PRIMARY OUTCOMES:
Ulcer area reduction rate | Pre-intervention, five weeks and ten weeks of treatment
  The ulcers will be measured with a paper ruler and photographed for later analysis of the images using the ImageJ program. The paper ruler will be positioned to measure the length and width of the ulcers.

SECONDARY OUTCOMES:
University of Texas Rankings | Pre-intervention, five weeks and ten weeks of treatment
  For analysis of ulcer depth, volunteers will be grouped into A1 and C1 (superficial ulcers), A2 and C2 (ulcers involving tendon or joint capsule) and A3 (ulcers involving bone).
Quality of life assessment | Pre-intervention, five weeks and ten weeks of treatment
  The EQ-5D tool will be used, consisting of five questions that assess the following aspects: mobility, personal care, usual activities, pain or discomfort, and anxiety/depression.
Glycemic level assessment | Once a week for ten weeks (20 sessions)
  Volunteers' blood glucose levels will be checked once a week throughout treatment.
Analysis of healing time and recurrence rate | Quarterly follow-up (3 months) after initial healing
  Healing time:Difference, in days, between the date of the first clinical record of the lesion and the date on which the wound is considered fully healed, characterized by complete epithelialization, absence of secretion and necrotic tissue.Recurrence: assessed based on the difference, in days, between the date of complete healing and the record of recurrence of the lesion in the same region, major amputation, death or the end of the study period.

IPD SHARING:
Plan to Share IPD: No